CLINICAL TRIAL: NCT02943343
Title: The China Pulmonary Thromboembolism Registry Study (CURES)
Brief Title: The China Pulmonary Thromboembolism Registry Study
Acronym: CURES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: 100 medical centers in the China PE-DVT network (Ambiguous)
Responsible Party: Principal Investigator, Zhenguo Zhai,MD,PhD, Ph.D, MD, Professor of Pulmonary and Critical Care Medicine, China-Japan Friendship Hospital
Other Study IDs: 2016YFC0905600
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Embolism; Deep Venous Thrombosis; Venous Thromboembolism
Keywords: Pulmonary embolism; Deep venous thrombosis; Venous thromboembolism; Registry; Real-world study
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Epidemiological data on pulmonary embolism (PE) in China needs to be updated and reported. The China Pulmonary Thromboembolism Registry Study (CURES) is designed to provide the cross-sectional spectrum and chronological trends of PE in China, as well as to reveal the intrinsic etiology and pathogenesis of the disease. The CURES is an ongoing large prospective multicenter registry, which was originally initiated in January 2009 via enrolling suspected or confirmed PE or PE with DVT (deep venous thrombosis) patients and assessed their in-hospital outcomes from 100 medical centers in the China PE-DVT network. As of July 2011, in order to determine the PE-relevant short-term outcomes, enrolled participants were followed-up for at least three months in a longitudinal manner. Since August 2016, with the launch and development of precision medicine research scheme in China, the main principle investigators of CURES decided to collect enrolled patients' blood samples with regular follow-ups every three or six months for at least two years (for long-term outcomes). The study protocol has been approved by the China-Japan Friendship Hospital ethics committee, and all collaborating centers received approvals from their local ethics committee. All patients provided written or verbal informed consent to their participation.

ELIGIBILITY:
Patients aged 18 years or above who are admitted to the 100 participating medical centers with suspected PE or PE with DVT are potentially eligible participants and consecutively enrolled in this registry.

Inclusion criteria:

* Objectively confirmed symptomatic PE or PE with DVT patients aged 18 years or above;
* Be able to provide written or verbal informed consent to participation.

Exclusion criteria:

* Younger than 18 years;
* Participation in a therapeutic clinical trial with an unknown drug;
* Inability for at least three-month follow-up since July 2011;
* Suspected PE or PE with DVT patients admitted to the hospital whereas without confirmed medical evidence;
* Patients with a history of PE or DVT readmitted to the hospital for examination or treatment however with no evidence of acute episode or recurrence;
* Withdrawal or lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic PE or PE with DVT are objectively confirmed by imaging tests. PE is confirmed by positive helical computed tomographic angiography of pulmonary artery (CTPA), high-probability ventilation-perfusion lung scintigraphy (V/Q), positive pulmonary angiography, or echocardiographic visualization of thrombus (in right atrium, right ventricle, pulmonary aorta trunk, or left/right pulmonary trunk), right atrium enlargement, or right ventricle hypokinesis while CTPA, V/Q scanning or pulmonary angiography are not applicable. DVT in the lower limbs is diagnosed with positive implications of compression ultrasonography (CUS) or computed tomographic venography (CTV).
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes at discharge | Two years
  Clinical outcomes at discharge or during hospitalization include disease recovery or cure, deterioration due to VTE or other comorbidities, and death (mainly all-cause and PE-specific mortality)
Other adverse events at discharge | Two years
  Other adverse events at discharge include bleeding (fatal bleeding, major bleeding, clinically relevant non-major bleeding), rash, liver dysfunction, thrombocytopenia, stroke or transient cerebral ischemia, myocardial infarction or acute coronary syndrome, etc.
Short-term (three months) and long-term (beyond three months and further forwards) clinical outcomes | Two years
  Clinical outcomes during short-term and long-term follow-ups include condition improvement or remission, recurrence of VTE (PE and DVT), chronic thromboembolic pulmonary hypertension (CTEPH), and death (mainly all-cause and PE-specific mortality)

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Zhai, Ph.D, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang D, Fan G, Lei J, Yang Y, Xu X, Ji Y, Yi Q, Chen H, Hu X, Liu Z, Mao Y, Zhang J, Shi J, Zhang Z, Wu S, Tao X, Xie W, Wan J, Zhang Y, Zhang S, Zhen K, Zhang Z, Fang B, Wang C, Zhai Z; China pUlmonary thromboembolism REgistry Study (CURES) investigators. LMWHs dosage and outcomes in acute pulmonary embolism with renal insufficiency, an analysis from a large real-world study. Thromb J. 2022 May 5;20(1):26. doi: 10.1186/s12959-022-00385-z. PMID 35513826
- [Derived] Zhai Z, Wang D, Lei J, Yang Y, Xu X, Ji Y, Yi Q, Chen H, Hu X, Liu Z, Mao Y, Zhang J, Shi J, Zhang Z, Wu S, Gao Q, Tao X, Xie W, Wan J, Zhang Y, Zhang S, Zhen K, Zhang Z, Fang B, Wang C; China pUlmonary thromboembolism REgistry Study (CURES) investigators. Trends in risk stratification, in-hospital management and mortality of patients with acute pulmonary embolism: an analysis from the China pUlmonary thromboembolism REgistry Study (CURES). Eur Respir J. 2021 Oct 28;58(4):2002963. doi: 10.1183/13993003.02963-2020. Print 2021 Oct. PMID 33986031
- [Derived] Lei J, Xu X, Ji Y, Yang Y, Yi Q, Chen H, Hu X, Liu Z, Mao Y, Zhang J, Shi J, Wang D, Zhang S, Zhang Z, Wu S, Gao Q, Tao X, Xie W, Wan J, Zhang Y, Zhang M, Shao X, Zhang Z, Fang B, Zhai Z, Wang C; China pUlmonary Thromboembolism REgistry Study (CURES) investigators. Rational and design of the China Pulmonary Thromboembolism Registry Study (CURES): A prospective multicenter registry. Int J Cardiol. 2020 Oct 1;316:242-248. doi: 10.1016/j.ijcard.2020.05.087. Epub 2020 Jun 6. PMID 32522676